CLINICAL TRIAL: NCT03622073
Title: Safety, Effectiveness and Acceptability of Misoprostol When Administered by Midwives Versus Physicians for Management of Incomplete Mid Trimester Abortion in Uganda: a Randomized Controlled Equivalence Trial.
Brief Title: Misoprostol Treatment of Mid Trimester Incomplete Abortion by Midwives and Doctors in Uganda.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: Karolinska Institutet (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC REF 2017-016
Record Dates: First submitted 2018-06-19; First posted 2018-08-09 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Incomplete Abortion
Keywords: Post abortion care; Misoprostol; Second trimester
MeSH Terms: conditions — Abortion, Incomplete

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Misoprostol treatment by Midwife (Experimental): Administration of misoprostol by the midwife and assessment for the primary outcome.
  Interventions: Other: Misoprostol treatment by Midwife
- Misoprostol treatment by Doctor (Active Comparator): Administration of misoprostol by the doctor and assessment for the primary outcome.
  Interventions: Other: Misoprostol treatment by Doctor

INTERVENTIONS:
Other: Misoprostol treatment by Midwife — Medical management of incomplete abortion
  Arms: Misoprostol treatment by Midwife
Other: Misoprostol treatment by Doctor — Medical management of incomplete abortion
  Arms: Misoprostol treatment by Doctor

SUMMARY:
It is estimated that 47,000 women die every year due to consequences of unsafe abortion globally. The majority of pregnancy related deaths occur in low income countries where induced abortion is restricted, unmet need for contraception is high, and women's status is low. Uganda has a high total fertility rate of 5.4 children per woman, low contraceptive prevalence rate of 39%, and more than half of these pregnancies are unintended. Induced abortion is controversial and restricted in Uganda and legally permitted only to save a woman's life. As a result, women often resort to unsafe abortion- that's either performed by a person lacking the necessary skills or in an environment that does not conform to minimal medical standards. Of the estimated 314,304 women who undergo unsafe abortions each year in Uganda, about 41% receive treatment for complications. This equates to an annual rate of 12 per 1,000 women aged 15-49 years being hospitalized for induced abortion complications, which is considered high in international comparison. In Uganda, outside the larger hospitals and private settings, access to safe post abortion care and surgical facilities are scarce. Studies have showed that trained midwives can deliver safe, effective and acceptable post abortion care using misoprostol in the first trimester. Currently in Uganda, treatment of second trimester incomplete abortion is restricted to physicians. This study will provide evidence on whether treatment for incomplete abortion using misoprostol by mid-level providers can be extended to the early second trimester period. The investigators hypothesize that misoprostol treatment for incomplete second trimester abortion provided by midwives is equivalent to that of physicians requiring no further surgical intervention. Women with incomplete abortion will be randomly allocated to undergo a clinical assessment and treatment with misoprostol either by physician or midwife with safety and effectiveness as main outcomes in the RCT carried out in hospital and high volume health centres in Central Uganda.

DETAILED DESCRIPTION:
This randomized controlled equivalence trial (RCT) implemented at eight hospitals and Health centres in Central Uganda will include 1192 eligible women with incomplete abortion of uterine size >12 weeks up to 18 weeks. Following informed consent, each participant will be randomly assigned to undergo a clinical assessment and treatment by either a midwife (intervention arm) or physician (control arm); receive 400mcg of misoprostol administered sublingually 3 hourly up to 5 doses within 24 hours at the health facility until a complete abortion is confirmed. Women who do not achieve a complete abortion within 24 hours will undergo a surgical method of uterine evacuation. Pre-discharge information on danger signs, contraceptive counselling and provision will be done with follow up 14 days later to assess secondary outcomes and acceptability. Analyses will be by Intention-to-Treat (ITT). Background characteristics and outcomes will be presented using descriptive statistics. Differences between groups will be analyzed using risk difference (95% CI) and equivalence established if it lies between the pre-defined range of -5% to +5%. Chi-square test will be used for comparison of outcome and t test used to compare mean values. P-values equal to or lower than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Vaginal bleeding
* With or without contractions with a uterine size > 12 weeks to < 18 weeks
* History of partial expulsion
* Open cervical os.

Exclusion Criteria:

* Known allergy to misoprostol,
* Unstable hemodynamic status (systolic blood pressure < 90mmHg) and shock
* Signs of pelvic infection and/or sepsis
* Previous caesarean delivery/uterine scar
* Suspected extra uterine pregnancy.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1191 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
Complete abortion | 24 hours from treatment initiation
  Number of participants who will have expelled all the products of conception as evidenced by cessation of abdominal cramps, vaginal bleeding and closed cervical os.

SECONDARY OUTCOMES:
Excessive vaginal bleeding | 24 hours from treatment initiation
  Participant reporting use of more than 3 pads in an hour.
Abdominal Pain | 24 hours from treatment initiation
  Pain will be defined as discomfort experienced in the lower abdomen using a visual analogue scale with a minimum score of zero representing no pain and a maximum score of 10 representing most pain. A higher score represents a worse outcome.
Unscheduled visits | 14-28 days post treatment
  Participant presenting at the study site when not expected
Women's acceptability of the post abortion care provider | 14-28 days post treatment
  Acceptability will be positive reporting of treatment experience, recommendation of method to a friend or reuse of same method.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina G Danielsson, PhD, Principal Investigator — Karolinska Institutet; Josaphat Byamugisha, PhD, Principal Investigator — Makerere University; Susan Atuhairwe, MD, Principal Investigator — Makerere University
Locations (14):
- Uganda (14):
  - Entebbe Hospital, Entebbe
  - Gombe Hospital, Gombe
  - Kawempe Hospital, Kampala
  - Kayunga Hospital, Kayunga
  - Kawolo Hospital, Lugazi
  - Luwero HC IV, Luwero
  - Masaka Hospital, Masaka
  - Mityana Hospital, Mityana
  - Mpigi HC IV, Mpigi
  - Kiganda HC IV, Mubende
  - Mukono HC IV, Mukono
  - Nakaseke Hospital, Nakaseke
  - Kasangati HC IV, Wakiso
  - Wakiso HC IV, Wakiso

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be available on request for systematic reviews. The particular data shared will depend on the request.
Time Frame: December 2025 to December 2030

REFERENCES:
- [Background] Faundes A. Strategies for the prevention of unsafe abortion. Int J Gynaecol Obstet. 2012 Oct;119 Suppl 1:S68-71. doi: 10.1016/j.ijgo.2012.03.021. Epub 2012 Aug 9. PMID 22883917
- [Background] Sedgh G, Bearak J, Singh S, Bankole A, Popinchalk A, Ganatra B, Rossier C, Gerdts C, Tuncalp O, Johnson BR Jr, Johnston HB, Alkema L. Abortion incidence between 1990 and 2014: global, regional, and subregional levels and trends. Lancet. 2016 Jul 16;388(10041):258-67. doi: 10.1016/S0140-6736(16)30380-4. Epub 2016 May 11. PMID 27179755
- [Background] Uganda Bureau of Statistcs (UBOS) and ICF. 2017. Uganda Demographic and Health Survey 2016: Key Indicators Report. Kampala, Uganda: UBOS, and Rockville, Maryland, USA: UBOS and ICF.
- [Background] Hussain R. Unintended pregnancy and abortion in Uganda. Issues Brief (Alan Guttmacher Inst). 2013 Jan;(2):1-8. PMID 23550324
- [Background] Prada E, Atuyambe LM, Blades NM, Bukenya JN, Orach CG, Bankole A. Incidence of Induced Abortion in Uganda, 2013: New Estimates Since 2003. PLoS One. 2016 Nov 1;11(11):e0165812. doi: 10.1371/journal.pone.0165812. eCollection 2016. PMID 27802338
- [Background] Mark AG, Edelman A, Borgatta L. Second-trimester postabortion care for ruptured membranes, fetal demise, and incomplete abortion. Int J Gynaecol Obstet. 2015 May;129(2):98-103. doi: 10.1016/j.ijgo.2014.11.011. Epub 2015 Jan 19. PMID 25660084
- [Background] Klingberg-Allvin M, Cleeve A, Atuhairwe S, Tumwesigye NM, Faxelid E, Byamugisha J, Gemzell-Danielsson K. Comparison of treatment of incomplete abortion with misoprostol by physicians and midwives at district level in Uganda: a randomised controlled equivalence trial. Lancet. 2015 Jun 13;385(9985):2392-8. doi: 10.1016/S0140-6736(14)61935-8. Epub 2015 Mar 27. PMID 25817472
- [Background] Cleeve A, Byamugisha J, Gemzell-Danielsson K, Mbona Tumwesigye N, Atuhairwe S, Faxelid E, Klingberg-Allvin M. Women's Acceptability of Misoprostol Treatment for Incomplete Abortion by Midwives and Physicians - Secondary Outcome Analysis from a Randomized Controlled Equivalence Trial at District Level in Uganda. PLoS One. 2016 Feb 12;11(2):e0149172. doi: 10.1371/journal.pone.0149172. eCollection 2016. PMID 26872219
- [Background] Moran M, Ortega J, Hodoglugil NN. Osur et al.'s Implementation of misoprostol for postabortion care in Kenya and Uganda: a qualitative evaluation. Glob Health Action. 2012 Jul 18;6:21786. doi: 10.3402/gha.v6i0.21786. No abstract available. PMID 23870184
- [Background] Pongsatha S, Tongsong T. Randomized controlled trial comparing efficacy between a vaginal misoprostol loading and non-loading dose regimen for second-trimester pregnancy termination. J Obstet Gynaecol Res. 2014 Jan;40(1):155-60. doi: 10.1111/jog.12147. Epub 2013 Sep 5. PMID 24033985
- [Background] Dawson AJ, Buchan J, Duffield C, Homer CS, Wijewardena K. Task shifting and sharing in maternal and reproductive health in low-income countries: a narrative synthesis of current evidence. Health Policy Plan. 2014 May;29(3):396-408. doi: 10.1093/heapol/czt026. Epub 2013 May 8. PMID 23656700
- [Background] Nabudere H, Asiimwe D, Mijumbi R. Task shifting in maternal and child health care: an evidence brief for Uganda. Int J Technol Assess Health Care. 2011 Apr;27(2):173-9. doi: 10.1017/S0266462311000055. Epub 2011 Mar 30. PMID 21450128
- [Derived] Atuhairwe S, Hanson C, Atuyambe L, Byamugisha J, Tumwesigye NM, Ssenyonga R, Gemzell-Danielsson K. Evaluating women's acceptability of treatment of incomplete second trimester abortion using misoprostol provided by midwives compared with physicians: a mixed methods study. BMC Womens Health. 2022 Nov 5;22(1):434. doi: 10.1186/s12905-022-02027-y. PMID 36335344
- [Derived] Atuhairwe S, Byamugisha J, Kakaire O, Hanson C, Cleeve A, Klingberg-Allvin M, Tumwesigye NM, Gemzell-Danielsson K. Comparison of the effectiveness and safety of treatment of incomplete second trimester abortion with misoprostol provided by midwives and physicians: a randomised, controlled, equivalence trial in Uganda. Lancet Glob Health. 2022 Oct;10(10):e1505-e1513. doi: 10.1016/S2214-109X(22)00312-6. Epub 2022 Aug 26. PMID 36030801
- [Derived] Atuhairwe S, Byamugisha J, Klingberg-Allvin M, Cleeve A, Hanson C, Tumwesigye NM, Kakaire O, Danielsson KG. Evaluating the safety, effectiveness and acceptability of treatment of incomplete second-trimester abortion using misoprostol provided by midwives compared with physicians: study protocol for a randomized controlled equivalence trial. Trials. 2019 Jun 21;20(1):376. doi: 10.1186/s13063-019-3490-5. PMID 31227019